

# PharmacoEpidemiology Group (PEG)

# Impact Evaluation of the Therapeutic Initiative's Uncomplicated Acute Cystitis Personalized Portrait and Therapeutics Letter

## **Analytic Protocol**

**Authors:** Greg Carney

**Creation date:** April 08, 2022

Last updated: Jan 31, 2023

Version: V 0.2

### Contents

| Introduction | 3 |
|---|---|
| Purpose | 3 |
| Study Purpose | |
| Research Question(s) / Hypothesis | 3 |
| Objectives | 4 |
| Methods | 4 |
| Study Dates: | 4 |
| Population (cohorts) | |
| Exposures | 7 |
| eferences | |
| | Purpose Study Purpose Research Question(s) / Hypothesis Objectives Methods Study Dates: Study Comparisons: Data sources. Population (cohorts) Exposures Medications Outcomes. Statistical Analysis Plan |

## **Document Control**

| Version | Date | Author(s) | Type of change |
|---------|-----------------|-----------|----------------------|
| 0.1 | April 08, 2022 | GC | First Draft |
| 0.2 | Jan 31, 2023 GC | | Minor clarifications |

**Study Name:** Impact Evaluation of the Therapeutic Initiative's Uncomplicated Acute Cystitis Personalized Portrait and Therapeutics Letter

Nickname: UTI Evaluation

Project Team: Greg Carney (Project lead) [Include role]

Anat Fisher (Clinical)

Malcolm Maclure (Methods)
Colin Dormuth (Methods)

Dana Stanley (Ethics/Coordinator)

**Data Access**: Health*ideas* including: ClaimsHist, MSP fee-for-service, hospital discharge abstracts, client roster, physician roster.

#### 1. Introduction

Indicators show that infections caused by antimicrobial resistant organisms continue to increase in Canada, and despite decades of antimicrobial stewardship programs the quality of antibiotic prescribing remains suboptimal. Continued efforts to preserve the effectiveness of antimicrobials to treat infectious diseases are essential, since misuse of antimicrobials is the primary mechanism driving resistance. V-Viii The treatment of cystitis is one indication where a change in antibiotic use was necessary. Uncomplicated acute cystitis (UAC) is the most prevalent form of urinary tract infection in women, and is most commonly caused by *escherichia coli* (E. coli). X, UAC is a common indication for antimicrobial treatment in healthy, non-pregnant women. Xi, Xii E. coli resistance to TMP-SMX and fluoroquinolones, historically the antibiotics most often used for UAC, has exceeded 20% in all areas of British Columbia, thus limiting the empirical effectiveness of these treatments. Due to increased resistance, Nitrofurantoin is now the best evidence supported treatment of infections caused by E. Coli or Staphylococcus Saprophyticus. Xiii

## 2. Purpose

#### Study Purpose

To conduct a randomized trial testing the effectiveness of personalized prescribing portraits and therapeutic letters on appropriate treatment for uncomplicated acute cystitis.

#### Research Question(s) / Hypothesis

Research Question: Determine the change in nitrofurantoin prescribing associated with the personal prescribing portrait and the therapeutics letter for UAC.

Hypothesis: The personal prescribing feedback portrait and the letter will each be associated with an increase in nitrofurantoin prescribing.

## 3. Objectives

To conduct a randomized trial testing the effectiveness of personalized prescribing portraits and therapeutic letters on appropriate treatment for uncomplicated acute cystitis.

#### 4. Methods

We conducted a randomized trial to analyze the effectiveness of a personalized prescribing portrait in the primary care setting in the province of British Columbia between September 2021 and March 2022.

Physicians are randomized to three groups:

| | Arm A | Arm B | Arm C |
|-----------------|------------------|------------|--------------|
| | ~33% | ~33% | ~33% |
| Initial mailing | Early Portrait + | | Early Letter |
| Sept 23, 2021 | Letter | Nothing | Only |
| | | Delayed | Delayed |
| Delayed mailing | | Portrait + | Portrait + |
| Mar 28, 2022 | | Letter | Letter |

<sup>\*</sup>Approximately 1,691 physicians were randomized to each group. However, not all will receive materials due to opt-outs and incorrect addresses.

#### Study Dates:

-Early mailing (groups A and C): 23-Sept-2021

-Delayed mailing (groups B and C): 28-Mar-2022

-Letter & Portrait topic released publicly on website: 28-Mar-2022

**Study Period**: September 24<sup>th</sup>, 2021 to March 28, 2022.

**Delay Period**: March 29, 2022 to Sept 28, 2022

#### Study Comparisons:

There will be four comparisons:

During the study period (Sept 23, 2021 to Mar 28, 2022):

- i. Arm A vs Arm B (impact of L+P combined)
- ii. Arm A vs Arm C (The added impact of P in physicians who received L)
- iii. Arm C vs Arm B (Impact of L)

During the study period (Sept 23, 2021 to Sept 28, 2022):

iv. Arm B vs Arm C (repeated messaging)



#### Data sources

B.C. Ministry of Health Health*ideas* data warehouse, including: ClaimsHist, MSP fee-for-service, hospital discharge abstracts, client roster, physician roster.

Estimated number of records/charts to be examined: 1691 physicians randomized to each group = 5,073. Estimate 6 UTI treated visits per physician = **30,438 patient records** to be included in the analysis.

#### Population (cohorts)

#### **Physicians:**

Physician eligibility criteria for randomization:

- i. Registered with the College of Physicians and Surgeons of B.C. (CPSBC)
- ii. Defined as a *General Practitioner* or *FP Emergency Medicine* according to the B.C. Ministry of Health's Medical Services Plan (MSP) with a license status of *private practice*, *temporary license*, *salaried*, *or post graduate*.
- iii. Valid mailing address in B.C according to the College of Physicians and Surgeons of British Columbia's public physician information.
- iv. Had >=100 prescriptions filled at a community pharmacy in 2020 according to PharmaNet claims.

Physician eligibility criteria to receive a prescribing portrait:

- i. Met the criteria for randomization above
- ii. Diagnosed >= 1 eligible patient with UAC in 2019 or 2020 (for delay group: 2020 to 2021

<sup>\*</sup>Approximately 1,691 physicians were randomized to each of the 3 study groups.

#### Patients:

Patient visits for UAC were identified from MSP billing records in which the first 3 digits of the ICD-9 diagnosis code in the record indicated 595 - Cystitis.

#### Include UTI codes:

- 1. 595, 595.0, 595.3-595.9 (cystitis) (but do not include 595.1, 595.2 chronic cystitis)
- 2. 599 or 599.0, 599.8, 599.9 UTI, site not specified (do not include if 599.1-599.7)
- 3. 788 or 788.9 or 788.1 symptoms involving urinary system or dysuria (do not include if 788.0, 788.2-788.8)
- 4. 596, 599.7, or 791

These UAC patients were then categorized according to whether they received antibiotic treatment on or within 5 days of the physician office visit recorded in the MSP billing record. Only count events where the diagnosing and prescribing physician are the same.

#### Patient exclusions:

- less than 77 days (2.5 months) MSP enrolment in the 91 days prior to visit
- Age <15 at time of UTI diagnosis</li>
- Male or missing sex
- Recurrent UTI:
  - A visit with a diagnosis of UTI in the prior 90 days, and/or
  - More than 4 visits in the 1095 days (3 years) before visit with a diagnosis of UTI
- Complicating factors:
  - Discharge from hospital in prior 30 days
  - Severe disease/infection of the kidney (pyelonephritis), ICD9: 590, 590.1, 590.2, 590.8, 590.9; ICD10: N10, N12, N15.1, N16 (within previous or following 10 days). Hospital admission or ED.
  - Indwelling catheter, based on ICD-9: V53.6, 996.64, 996.76, 996.31.
     ICD10: T83.0x, Z46.6, Z96.0, in 91 days prior to UTI diagnosis
  - Impaired renal function, fee item: 33758, 33723, 33759, 33761 or if they have a visit with a nephrologist (prior 365 days)
  - Structural and functional abnormality of urinary tract (prior 365 days)
     [ICD9: 16.9, 137.2, 997.5, 939.3, 939.9, 947.4, V130 ICD10: A181, B901,
     N998, N999, T198, T199, T283, T288, Z874.]
  - Pregnant women, fee item: 14090, 14091, 36360, 36361, 04717 codes or ICD 646.6, V22.x, V23.x in the 270 days before the UTI visits + no record of pregnancy outcome after pregnancy code and before UTI event (ICD9 630.x, 631.x, 632.x, 633.x, 634.x, 635.x, 636.x, 637.x, V24.x, V27.x, 656.4 or ICD10 000.x, 001.x, 002.x, 003.x, 004.x, 005.x, Z37.x, 036.4x)

- Diagnosis of STI within 14 days before or after UTI visit (ICD9: 090-099, ICD10: A50-A64)
- Chronic Kidney Disease (ICD9: 585.x, ICD10: N18) MSP complex care code: N585, R585, I585, H585, D585, C585, K573) in previous 365 days
- Physician visit where patient had any oral, intravenous, or injection antibiotics (ATC: J01) in previous 91 days dispensed by any physician
- Patients with a dispensation under Plan P or B (on abx fill date or within 3 months after)

#### Exposures

Female patient visits for UAC identified from physician MSP billing records in which the first 3 digits of the ICD-9 diagnosis code in the record indicated *595 – Cystitis*.

#### Medications

All oral formulation prescription antibiotics available in BC were included in the portrait.

Nitrofurantoin identified using ATC: J01XE01

#### Outcomes

The primary outcome is the incidence of women treated with nitrofurantoin in the 5-day period following a diagnosis of Uncomplicated Acute Cystitis, including the day of diagnosis.

## 5. Statistical Analysis Plan

- 1. **Baseline Characteristics:** Physicians and Patients by Study Group. Age (mean, sd), age groups, sex, urban vs rural.
- 2. **Trends:** Weekly prescribing line chart by randomized physician group of Nitrofurantoin, Ciprofloxacin, and TMP-SMX, from 6 months prior to first mailing to the end of the delay period 6 months after the delayed mailing (September 2022). This will illustrate background trends in prescribing patterns.
- 3. **Relative Risk:** Prescribing in the early and delayed intervention groups will be compared 6 months pre/post intervention. A 4-way comparison of numerators during the pre/post periods between the early and delay groups will provide an odds ratio that approximates the relative risk. xiv,xv Do this for each of the four study comparisons listed in Section 4.

| Acute cystitis episodes = n | | Intervention Physicians | | | Del | Delayed Contol Physicians | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Expected | | Time Period | | | Time Period | | | Crude | Adjusted | 95% CL | |
| Outcome Measures | Change | <u>Pre</u> | | Post | | <u>Pre</u> | | Post | | OR | OR |
| | | YES | NO | YES | NO | YES | NO | YES | NO | | |
| Nitrofurantoin | + | a | b | С | d | е | f | g | h | | |
| Ciprofloxacin | - | | | | | | | | | | |
| TMP_SMX | - | | | | | | | | | | |
| Other | - | | | | | | | | | | |
| No Treatment | n/c | | | | | | | | | | |

Crude OR = 
$$\frac{(c * h)}{(g * d)}$$

Evaluation is a 4-way comparison: the ratio of change in the early group between pre and post intervention is compared to the same ratio of change in the delayed group.

Adjusted OR = 
$$\frac{\text{Crude OR}}{(a * f)}$$
10 
$$(e * b)$$

#### References:

- Maclure 2006. Measuring prescribing improvements in pragmatic trials of educational tools for general practitioners. *Basic Clin Pharmacol Toxicol*.
- 2. Dormuth 2012. A randomized trial assessing the impact of a personalized feedback portrait on statin prescribing in primary care. J Contin Educ Health Prof.

#### References

<sup>1</sup> Public Health Agency of Canada . 2020. Canadian antimicrobial resistance surveillance system report – update 2020. <a href="https://www.canada.ca/en/public-health/services/publications/drugs-health-products/canadian-antimicrobial-resistance-surveillance-system-2020-report.html">https://www.canada.ca/en/public-health/services/publications/drugs-health-products/canadian-antimicrobial-resistance-surveillance-system-2020-report.html</a>. Accessed Nov 30, 2021.

- <sup>II</sup> Saatchi A, Yoo JW, Schwartz KL, Silverman M, Morris AM, Patrick DM, McCormack J, Marra F. Quantifying the Gap between Expected and Actual Rates of Antibiotic Prescribing in British Columbia, Canada. Antibiotics (Basel). 2021 Nov 22;10(11):1428. doi: 10.3390/antibiotics10111428. PMID: 34827366; PMCID: PMC8615253.
- McCubbin KD, Anholt RM, de Jong E, Ida JA, Nóbrega DB, Kastelic JP, Conly JM, Götte M, McAllister TA, Orsel K, Lewis I, Jackson L, Plastow G, Wieden HJ, McCoy K, Leslie M, Robinson JL, Hardcastle L, Hollis A, Ashbolt NJ, Checkley S, Tyrrell GJ, Buret AG, Rennert-May E, Goddard E, Otto SJG, Barkema HW. Knowledge Gaps in the Understanding of Antimicrobial Resistance in Canada. Front Public Health. 2021 Oct 20;9:726484. doi: 10.3389/fpubh.2021.726484. PMID: 34778169; PMCID: PMC8582488.
- <sup>iv</sup> Saatchi A, Morris AM, Patrick DM, Mccormack J, Reyes RC, Morehouse P, Reid J, Shariff S, Povitz M, Silverman M, Marra F. Outpatient antibiotic use in British Columbia, Canada: reviewing major trends since 2000. JAC Antimicrob Resist. 2021 Aug 12;3(3):dlab116. doi: 10.1093/jacamr/dlab116. PMID: 34396123; PMCID: PMC8360297.
- <sup>v</sup> Davies J, Davies D. Origins and evolution of antibiotic resistance. Microbiol Mol Biol Rev. 2010 Sep;74(3):417-33. doi: 10.1128/MMBR.00016-10. PMID: 20805405; PMCID: PMC2937522.<sup>vi</sup> Ruckert A, Fafard P, Hindmarch S, Morris A, Packer C, Patrick D, Weese S, Wilson K, Wong A, Labonté R. Governing antimicrobial resistance: a narrative review of global governance mechanisms. J Public Health Policy. 2020 Dec;41(4):515-528. doi: 10.1057/s41271-020-00248-9. PMID: 32908184; PMCID: PMC7479750.
- vii Paphitou NI. Antimicrobial resistance: action to combat the rising microbial challenges. Int J Antimicrob Agents. 2013 Jun;42 Suppl:S25-8. doi: 10.1016/j.ijantimicag.2013.04.007. Epub 2013 May 16. PMID: 23684003.
- viii Rudnick W, Science M, Thirion DJG, Abdesselam K, Choi KB, Pelude L, Amaratunga K, Comeau JL, Dalton B, Delport J, Dhami R, Embree J, Émond Y, Evans G, Frenette C, Fryters S, German G, Grant JM, Happe J, Katz K, Kibsey P, Kosar J, Langley JM, Lee BE, Lefebvre MA, Leis JA, McGeer A, Neville HL, Simor A, Slayter K, Suh KN, Tse-Chang A, Weiss K, Conly J; Canadian Nosocomial Infection Surveillance Program. Antimicrobial use among adult inpatients at hospital sites within the Canadian Nosocomial Infection Surveillance Program: 2009 to 2016. Antimicrob Resist Infect Control. 2020 Feb 13;9(1):32. doi: 10.1186/s13756-020-0684-2. PMID: 32054539; PMCID: PMC7020554.
- <sup>ix</sup> Li R, Leslie SW. Cystitis. 2021 Feb 10. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2021 Jan–. PMID: 29494042.
- \* Lala V, Minter DA. Acute Cystitis. 2020 Nov 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2021 Jan–. PMID: 29083726.
- xi Kang CI, Kim J, Park DW, Kim BN, Ha US, Lee SJ, Yeo JK, Min SK, Lee H, Wie SH. Clinical Practice Guidelines for the Antibiotic Treatment of Community-Acquired Urinary Tract Infections. Infect Chemother. 2018 Mar;50(1):67-100. doi: 10.3947/ic.2018.50.1.67. PMID: 29637759; PMCID: PMC5895837. xii Gupta K, Hooton TM, Naber KG, Wullt B, Colgan R, Miller LG, Moran GJ, Nicolle LE, Raz R, Schaeffer AJ, Soper DE; Infectious Diseases Society of America; European Society for Microbiology and Infectious Diseases. International clinical practice guidelines for the treatment of acute uncomplicated cystitis and pyelonephritis in women: A 2010 update by the Infectious Diseases Society of America and the European Society for Microbiology and Infectious Diseases. Clin Infect Dis. 2011 Mar 1;52(5):e103-20. doi: 10.1093/cid/ciq257. PMID: 21292654.

xiii Gupta K. et al. Short-Course Nitrofurantoin for the Treatment of Acute Uncomplicated Cystitis in Women. Arch Intern Med. 2007;167(20):2207-2212.

xiv Maclure M, Nguyen A, Carney G, Dormuth C, Roelants H, Ho K, Schneeweiss S. Measuring prescribing improvements in pragmatic trials of educational tools for general practitioners. Basic Clin Pharmacol Toxicol. 2006 Mar;98(3):243-52. doi: 10.1111/j.1742-7843.2006.pto\_301.x. PMID: 16611198.

<sup>&</sup>lt;sup>xv</sup> Dormuth CR, Carney G, Taylor S, Bassett K, Maclure M. A randomized trial assessing the impact of a personal printed feedback portrait on statin prescribing in primary care. J Contin Educ Health Prof. 2012 Summer;32(3):153-62. doi: 10.1002/chp.21140. PMID: 23008077.